CLINICAL TRIAL: NCT00003910
Title: A Phase II Study of Initial Treatment With Methotrexate in Large Granular Lymphocytic (LGL) Leukemia
Brief Title: Methotrexate With or Without Cyclophosphamide in Treating Patients With Lymphocytic Leukemia
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000067089; U10CA021115 (NIH); E5998 (Other: ECOG)
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Results first posted 2013-05-27 (Estimated); Last update posted 2023-07-05 (Actual); Status verified 2023-06

CONDITIONS: Leukemia
Keywords: stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; stage IV chronic lymphocytic leukemia; T-cell large granular lymphocyte leukemia; LGL clone
MeSH Terms: conditions — Leukemia; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Large Granular Lymphocytic | interventions — Cyclophosphamide; Methotrexate; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Methotrexate (Cy if no response to MTX) (Experimental): MTX given orally at 10 mg/m2 in divided doses once weekly. Prednisone was given orally at 1 mg/kg per day for 30 days and then tapered off in the subsequent 24 days. Patients not responding to MTX after 4 months received Cy orally at 100 mg daily in step two with the same prednisone schedule.
  Interventions: Drug: Cyclophosphamide; Drug: Methotrexate; Drug: Prednisone

INTERVENTIONS:
Drug: Cyclophosphamide — Patients not responding to MTX after 4 months received Cy orally at 100 mg daily in step two with the same prednisone schedule. In patients showing a partial response, but not a CR, the maximum period of therapy was 1 year.
Drug: Methotrexate — Initial treatment consisted of MTX given orally at 10 mg/m2 in divided doses once weekly.
Drug: Prednisone — Prednisone was given orally at 1 mg/kg per day for 30 days and then tapered off in the subsequent 24 days.

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of methotrexate with or without cyclophosphamide in treating patients who have lymphocytic leukemia with neutropenia or anemia.

DETAILED DESCRIPTION:
LGL leukemia is characterized by clonal expansion of cytotoxic T cells. Prominent clinical features include neutropenia, anemia, and rheumatoid arthritis. The terminal effector memory phenotype (CD3+/CD8+/CD57+/CD45RA+/CD62L-) of leukemic LGL suggest a pivotal chronic antigen driven immune response. LGL survival is then promoted by PDGF and IL-15, resulting in global dysregulation of apoptosis and resistance to normal pathways of activation-induced death. These pathogenic features explain why treatment of LGL leukemia is based on immunosuppression therapy. However, no standard therapy has been established due to the absence of large prospective trials.

Oral low dose MTX has been shown to be efficacious in the treatment of neutropenia. However, response to MTX is slow, requiring several months for the neutrophil count to increase above 500/mm3. Also, complete clinical remission may not be achieved until after one year of MTX therapy. Oral Cy has been the primary drug used for the treatment of severe transfusion-dependent anemia. Beneficial clinical effects are seen despite this treatment having no apparent effect on the abnormal LGL clone. Normal hematocrits are maintained after cessation of Cy and these results contrast the effects seen with MTX, in which clinical remissions are often associated with the disappearance of the clone.

This phase II trial undertaken by the Eastern Cooperative Group (ECOG) was initiated to investigate the mechanism of treatment response in patients with LGL leukemia, who need treatment for anemia or neutropenia.

ELIGIBILITY:
Inclusion:

* Phenotypic studies from peripheral blood showing CD3+, CD57+ cells greater than 400/mm3 or CD8+ cells greater than 650/mm3 within eight weeks prior to registration
* Evidence for clonal T-cell receptor gene rearrangement within one year prior to registration
* At least one of the following: Severe neutropenia less than 500/mm3, neutropenia associated with recurrent infections, symptomatic anemia, or transfusion-dependent anemia
* Bilirubin ≤ 2.0 mg/dl, SGOT(AST) ≤ 1.5 times normal, and Creatinine ≤ 2.0 mg/dl within 4 weeks prior to registration
* ECOG performance status of 0-2
* At least 18 years of age
* Written informed consent

Exclusion:

* Prior therapy with oral MTX or oral Cy
* Previous or concurrent malignancies except inactive non-melanoma skin cancer, in situ carcinoma of the cervix, or other cancer if the patient has been disease free for over 5 years
* Pregnant or breast-feeding for female patients
* Serious medical illness, other than that treated by the study, which would limit survival to less than 2 years, or psychiatric condition which would prevent informed consent

Note: to be eligible for step 2 of this study, patients were required to have no response after at least 4 months of methotrexate treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 1999-09-15 (Actual); Primary Completion 2010-12-01 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas P. Loughran, MD, Study Chair — Milton S. Hershey Medical Center
Locations (68):
- United States (68):
  - Aurora Presbyterian Hospital, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose Cancer Center at Penrose Hospital, Colorado Springs, Colorado
  - St. Anthony Central Hospital, Denver, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - St. Joseph Hospital, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - CCOP - Colorado Cancer Research Program, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - St. Mary's Regional Cancer Center at St. Mary's Hospital and Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Hope Cancer Care Center at Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - St. Mary - Corwin Regional Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Medical Center of Central Georgia, Macon, Georgia
  - Rush-Copley Cancer Care Center, Aurora, Illinois
  - Robert H. Lurie Comprehensive Cancer Center at Northwestern University, Chicago, Illinois
  - Evanston Northwestern Healthcare - Evanston Hospital, Evanston, Illinois
  - Joliet Oncology-Hematology Associates, Limited - West, Joliet, Illinois
  - North Shore Oncology and Hematology Associates, Limited - Libertyville, Libertyville, Illinois
  - Carle Cancer Center at Carle Foundation Hospital, Urbana, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - Methodist Cancer Center at Methodist Hospital, Indianapolis, Indiana
  - Saint Anthony Memorial Health Centers, Michigan City, Indiana
  - McFarland Clinic, PC, Ames, Iowa
  - Mercy Cancer Center at Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Hematology-Oncology Associates, LLP, Sioux City, Iowa
  - Mercy Medical Center - Sioux City, Sioux City, Iowa
  - St. Luke's Regional Medical Center, Sioux City, Iowa
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy and Unity Cancer Center at Mercy Hospital, Coon Rapids, Minnesota
  - Fairview Southdale Hospital, Edina, Minnesota
  - Mercy and Unity Cancer Center at Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - HealthEast Cancer Care at St. John's Hospital, Maplewood, Minnesota
  - Minnesota Oncology Hematology, PA - Maplewood, Maplewood, Minnesota
  - Virginia Piper Cancer Institute at Abbott - Northwestern Hospital, Minneapolis, Minnesota
  - Hennepin County Medical Center - Minneapolis, Minneapolis, Minnesota
  - Hubert H. Humphrey Cancer Center at North Memorial Outpatient Center, Robbinsdale, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Park Nicollet Cancer Center, Saint Louis Park, Minnesota
  - Regions Hospital Cancer Care Center, Saint Paul, Minnesota
  - HealthEast Cancer Care at St. Joseph's Hospital, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - St. Francis Cancer Center at St. Francis Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - HealthEast Cancer Care at Woodwinds Health Campus, Woodbury, Minnesota
  - Minnesota Oncology Hematology, PA - Woodbury, Woodbury, Minnesota
  - Aultman Cancer Center at Aultman Hospital, Canton, Ohio
  - St. Rita's Medical Center, Lima, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Central Pennsylvania Hematology and Medical Oncology Associates, PC, Lemoyne, Pennsylvania
  - Lewistown Hospital, Lewistown, Pennsylvania
  - Fox Chase Cancer Center - Philadelphia, Philadelphia, Pennsylvania
  - McGlinn Family Regional Cancer Center at Reading Hospital and Medical Center, Reading, Pennsylvania
  - Mount Nittany Medical Center, State College, Pennsylvania
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Froedtert Hospital and Medical College of Wisconsin, Milwaukee, Wisconsin
  - Medical College of Wisconsin Cancer Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study accrued 59 patients between July 16, 1999 and March 24, 2009. The first patient was accrued on September 15, 1999. The study terminated with 59 patients on March 24, 2009 due to slower than expected accrual.
Groups:
- Methotrexate: MTX given orally at 10 mg/m2 in divided doses once weekly. Prednisone was given orally at 1 mg/kg per day for 30 days and then tapered off in the subsequent 24 days. If patient had a partial response, MTX was continued for up to 1 year. If patient had CR, MTX was continued for 1 month.
  If no response, then pt went onto step 2 and received CY.
- Cyclophosphomide: Patients not responding to MTX after 4 months received Cy orally at 100 mg daily in step two with the same prednisone schedule.
Period: Step 1
Arm/Group | Methotrexate | Cyclophosphomide
Started | 55 (Of 59 (step 1), 4 pts were ineligible.) | 0
Completed | 55 | 0
Not Completed | 0 | 0
Period: Step 2
Arm/Group | Methotrexate | Cyclophosphomide
Started | 0 | 16 (The 16 includes 2 ineligible pts.)
Completed | 0 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Methotrexate: MTX given orally at 10 mg/m2 in divided doses once weekly. Prednisone was given orally at 1 mg/kg per day for 30 days and then tapered off in the subsequent 24 days. Patients not responding to MTX after 4 months received Cy orally at 100 mg daily in step two with the same prednisone schedule.
Arm/Group | Methotrexate
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.4 (17.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 30
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Complete or Partial Response to Treatment With MTX
Description: We will report the overall response rate below. Complete remission requires that all of the following be present for at least four weeks: The patient must have a normal CBC including neutrophil count > 1500/mm3, lymphocyte count< 4000/mm3, hemoglobin > 11 g/dl, and platelet count > 100,000/mm3. In addition, the patient must have a normal LGL count. A complete response will be attained if CD8+ cells were less than 760/mm³. A partial response will be defined as achievement of any one of the following in the absence of CR. The response must last for at least four weeks:In patients being treated for severe neutropenia (less than 500 neutrophils/mm3) an improvement to over 500 neutrophils/mm3 will be considered a partial response, as long as that improvement represents at least a 50% improvement.
Time Frame: Assessed during the first 4 months, then at least every three months for two years. Then every six months until five years after study entry, and every 12 months thereafter until full study stop date.
Population: Of the 59 pts, 4 were ineligible and excluded from the analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Methotrexate
Number analyzed (Participants) | 55
proportion of participants | 0.39 [0.26 to 0.53]

2. Secondary Outcome: Proportion of Patients With Complete or Partial Response to Treatment of CY Among Patients Failing to Respond to MTX
Description: as for outcome 1
Time Frame: Assessed during the first 4 months of treatment and followed until reaching full study stop date
Population: Eligible patients who received Cy after failing to respond to MTX are included in this analysis.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Cyclophosphamide (Cy): Patients not responding to MTX after 4 months received Cy orally at 100 mg daily in step two with the same prednisone schedule. In patients showing a partial response, but not a CR, the maximum period of therapy was 1 year.
Arm/Group | Cyclophosphamide (Cy)
Number analyzed (Participants) | 14
proportion of participants | 0.64 [0.35 to 0.87]

ADVERSE EVENTS:
Time Frame: Assessed every 30 days while on treatment and for 30 days after the end of treatment.
Description: Here we look at all patients, all 59, whereas we excluded the ineligible patients from the baseline tables etc (n=55) as is standard to do in our final reports for ECOG.
Groups:
- Cyclophosphamide: step 2 patients who received CY
Arm/Group | Methotrexate | Cyclophosphamide
Serious Adverse Events (participants affected / at risk) | 56/59 | 8/16
Other Adverse Events (participants affected / at risk) | 56/59 | 6/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=59) | Cyclophosphamide (N=16)
Anemia (Blood and lymphatic system disorders) | 13 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Cough (General disorders) | 1 | 0
Creatinine (Blood and lymphatic system disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Fatigue (General disorders) | 5 | 0
Hemmorhage (Blood and lymphatic system disorders) | 1 | 0
Hyperglycemia (Blood and lymphatic system disorders) | 6 | 2
Hypertension (Cardiac disorders) | 1 | 0
Hyponatremia (Metabolism and nutrition disorders) | 2 | 0
Hypoxia (Metabolism and nutrition disorders) | 2 | 0
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 6 | 0
Infection without neutropenia (Infections and infestations) | 3 | 0
Leukopenia (Blood and lymphatic system disorders) | 10 | 6
Lymphopenia (Blood and lymphatic system disorders) | 5 | 7
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 30 | 6
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 5 | 1
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 6 | 1
Melena/GI bleeding (Gastrointestinal disorders) | 0 | 1
Depressed level of consciousness (Psychiatric disorders) | 0 | 1
Cardiac-left ventricular function (Cardiac disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hematuria (Renal and urinary disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=59) | Cyclophosphamide (N=16)
AST increased (Metabolism and nutrition disorders) | 21 | 0
Alkaline Phosphatase Increased (Metabolism and nutrition disorders) | 9 | 0
Anemia (Blood and lymphatic system disorders) | 41 | 5
Anorexia (Metabolism and nutrition disorders) | 11 | 0
Bilirubin Increased (Metabolism and nutrition disorders) | 15 | 0
Constipation (Gastrointestinal disorders) | 4 | 0
Creatinine (Metabolism and nutrition disorders) | 11 | 0
Diarrhea (Gastrointestinal disorders) | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 11 | 1
Edema (Metabolism and nutrition disorders) | 5 | 0
Fatigue (General disorders) | 34 | 0
Fever (General disorders) | 8 | 0
Hyperglycemia (Metabolism and nutrition disorders) | 34 | 3
Hypoalemia (Metabolism and nutrition disorders) | 9 | 0
Hypoglycemia (Metabolism and nutrition disorders) | 7 | 0
Hypokalemia (Metabolism and nutrition disorders) | 9 | 0
Hyponatremia (Metabolism and nutrition disorders) | 14 | 0
Infection with grade 3 or 4 neutropenia (Infections and infestations) | 7 | 0
Insomnia (General disorders) | 10 | 0
Leukopenia (Blood and lymphatic system disorders) | 37 | 6
Nausea (Gastrointestinal disorders) | 14 | 0
Neutropenia (Blood and lymphatic system disorders) | 49 | 6
Stomatitis (Gastrointestinal disorders) | 10 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 20 | 1
Cardiac-left ventricular function (Cardiac disorders) | 0 | 1
Melena/GI bleeding (Gastrointestinal disorders) | 0 | 1
Depressed level of consciousness (Psychiatric disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Infection with unknown ANC (Infections and infestations) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No